CLINICAL TRIAL: NCT02902081
Title: Effects of Cannabidiol on Responses to Emotional Stimuli
Brief Title: Cannabidiol and Emotional Stimuli
Acronym: CAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB13-0215
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-04

CONDITIONS: Drug Addiction
MeSH Terms: conditions — Substance-Related Disorders | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Oral placebo administered once prior to subjective drug effects questionnaires and behavioral tasks.
  Interventions: Drug: Placebo
- Cannabidiol (Experimental): (300 mg, 600 mg, 900 mg) cannabidiol administered once prior to subjective drug effects questionnaires and behavioral tasks.
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol
  Arms: Cannabidiol
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this research is to examine the effect of cannabidiol (CBD), a cannabinoid compound found in marijuana, on responses to emotional stimuli. Both preclinical and clinical studies indicate that CBD may act to reduce anxiety without excessive sedative side-effects. Thus the investigators hypothesize that CBD may reduce responses specifically to negative emotional and social stimuli, including pictures and emotional faces, without altering responses to positive stimuli. To examine this, the investigators will administer placebo, 300mg, 600mg, and 900mg CBD to healthy normal adults in a double-blind within-subjects study. The investigators will measure subjective and subtle physical responses to positive and negative stimuli using measures that have been characterized with classic anxiety-reducing drugs and drugs of abuse. Further, the investigators will examine whether CBD-induced changes in these measures of emotional response relate to changes in actual behavior in a controlled social interaction. These results will allow the investigators to examine the potential usefulness of CBD as an anxiety-reducing drug, and suggest mechanisms by which CBD may reduce anxiety.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years of age.
* 38 healthy volunteers (19 male, 19 female; age range 18-35 years)
* All participants recruited without regard to race, religion or ethnicity through posters, advertisements and word-of-mouth referrals.
* Candidates screened in accordance with our general screening protocol, approved by the IRB under Protocol #13681B, which includes a physical, EKG, psychiatric screening interview and detailed drug use history questionnaire.

Exclusion Criteria:

* Individuals with a medical condition contraindicating study participation, as determined by the study site physician.
* Individuals regularly using any medications aside from hormonal contraception in women.
* Individuals with a current (active in the past year) DSM-IV Axis I mood, anxiety, eating, or substance dependence disorder or a lifetime history of a psychotic disorder or mania.
* Women who are pregnant, nursing, or planning to become pregnant in the next 3 months
* Participants reporting a known or suspected allergy to cannabinoids.
* The self-report questionnaires the investigators use require fluency in English, and have not been translated and validated in other languages, thus individuals with less than a high-school education or those not fluent in English were excluded, as lack of English familiarity at a high school level may compromise our ability to interpret their self-reports.
* Individuals with a BMI below 19 or above 30, as this would change dosing requirements.
* Individuals who report using marijuana >100 times in their lifetime, to reduce variation in possible developed tolerance to CBD.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2013-02; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- ALL Study Participants: This is a within-subjects study design in which "all" participants received "all" three does (300, 600, and 900 mg oral) of cannabidol and a placebo in randomized order.
Period: Overall Study
Arm/Group | ALL Study Participants
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ALL Study Participants
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 22
  African-American | 10
  Other | 6

OUTCOME MEASURES:

1. Primary Outcome: Positivity Ratings of Social Images
Description: Using the International Affective Picture System (IAPS; Lang et al. 1999), participants viewed standardized positive, negative and neutral pictures from the IAPS. The negative and positive images were matched on degree of valence and arousal. An Evaluative Space Grid rating followed each picture to collect subjective reactions. Ratings are on a 9-pt scale. The range of the scale is from 1 to 9 (Min score 1, max score 9). The total score is reported. Higher numbers represent more positive valence or greater arousal. Drug treatment: within-subjects; every participant received all drug doses, counter-balanced.
Time Frame: End of study (time 0 and approximately 4 weeks later), week 4 reported.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Placebo: Placebo capsule administered once prior to subjective drug effects questionnaires and behavioral tasks.
- 300 mg Cannabidiol: (300 mg) cannabidiol administered once prior to subjective drug effects questionnaires and behavioral tasks.
- 600 mg Cannabidiol: (600 mg) cannabidiol administered once prior to subjective drug effects questionnaires and behavioral tasks.
- 900 mg Cannabidiol: (900 mg) cannabidiol administered once prior to subjective drug effects questionnaires and behavioral tasks.
Arm/Group | Placebo | 300 mg Cannabidiol | 600 mg Cannabidiol | 900 mg Cannabidiol
Number analyzed (Participants) | 38 | 38 | 38 | 38
score on a scale
  Positive Image | 1.96 (0.11) | 1.68 (0.13) | 1.86 (0.10) | 1.93 (0.11)
  Negative Image | 0.47 (0.07) | 0.48 (0.08) | 0.41 (0.06) | 0.35 (0.06)
  Neutral Image | 1.12 (0.10) | 0.99 (0.10) | 1.08 (0.08) | 1.13 (0.10)

ADVERSE EVENTS:
Time Frame: .Through study completion, an average of 5 weeks.
Groups:
- Placebo: Oral placebo administered once prior to subjective drug effects questionnaires and behavioral tasks.
  Placebo
Arm/Group | Placebo | Cannabidiol
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT02902081/Prot_SAP_000.pdf